CLINICAL TRIAL: NCT05429242
Title: Placental Thickness and Pregnancy Outcomes
Brief Title: The Relation Between Placental Volume at the 1st Trimester and Perinatal Prognosis
Status: Completed | Type: Observational
Sponsor: Siirt University (Other)
Responsible Party: Principal Investigator, Serif Aksin, associate professor, Siirt University
Other Study IDs: SiirtUNIV
Record Dates: First submitted 2022-06-11; First posted 2022-06-23 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Pregnancy Complications; Perinatal Problems; Maternal-Fetal Relations
Keywords: placental volume; perinatal prognosis; first trimester; pregnancy
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ultrasonographic examination — Measurement of placental volume at the first trimester of pregnancy by using ultrasound.

SUMMARY:
It has been known for years that placental transport and endocrine and metabolic functions of the placenta are the main determinants of fetal nutrition and homeostasis. And placental capacity is roughly related to the weight of this organ. It has long been understood that placental weight at birth is also positively associated with birth weight. Since the 1970s, it has been possible to assess the size of the placenta in early pregnancy using two-dimensional (2D) ultrasonography (USG). Since then, it has been estimated that placental size is associated with fetal development. However, the difficulty in defining the required sonographic planes due to the technology of that time-limited the usefulness of this technique. As studies on this subject increase with the development of technology, it has now been shown that low placental volume at 11-13 weeks is associated with babies small for gestational age (SGA), fetal growth restriction, and preeclampsia. Pregnancy complications place a severe burden on the health system. Detection of these complications in the early period will prevent maternal and fetal mortality and morbidity. A relationship that predicts obstetric, fetal, and perinatal risks with placental thickness and width measurement with USG, a non-invasive method, in an early period such as the 1st trimester, will enable a proactive approach to complications. In our study, the investigators plan to present the perinatal results they obtained rather than investigating a specific relationship. The investigators think that the results of their study will make a profound contribution to the literature.

DETAILED DESCRIPTION:
This study aims to determine the relationship between the calculated placental volume in the 1st trimester and poor perinatal outcomes. For this purpose, approximately 360 pregnant women, who were followed up in Siirt Training and Research Hospital between June 2022 and June 2023 and were in their first trimester of pregnancy, will be included in the study. The pregnant woman's age, pregnancy history, and medical history will be recorded. The patient's gestational week, placental volume, and location will be recorded during the examination. All participants will be followed up until delivery. During delivery, gestational week, delivery type, fetal weight, APGAR score, baby gender, and pregnancy outcomes, preeclampsia, Gestational Diabetes, Gestational Hypertensive diseases, Premature rupture of membranes, preterm labor, oligohydramnios, polyhydramnios, presentation anomaly, Intrauterine death, Perinatal fetal disorders such as distress, intrauterine growth retardation, preeclampsia, placental abruption, placental invasion anomaly, placental implantation anomalies, postmaturity will be recorded. In the light of the information gathered, the relationship between placental volume in the 1st trimester and perinatal prognosis will be determined.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* 1.st trimester pregnancy

Exclusion Criteria:

* history of chronic hypertension
* history of pre gestational diabetes
* history of chronic diseases
* excessive consumption of alcohol
* smoking pregnants
* kidney disorders

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women over the age of 18 and at 11-14 weeks of pregnancy
Sampling Method: Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2022-06-11 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Placental thickness in millimetres and pregnancy outcomes | From the 1.st trimester of pregnancy up to the first month after birth ( the perinatal period,(( about 7 months ))
  The relationship between placental volume in the 1st trimester and perinatal prognosis will be tried to be determined.
Pregnancy outcomes | Pregnancy Week at the time of birth from the first three -month period of pregnancy (about 7 months)
  Gestational age in weeks during delivery
Pregnancy outcomes | Fetal weight at the time of birth from the first three -month period of pregnancy (about 7 months)
  Fetal weight in grams
Pregnancy outcomes | At the first minute and 5th minute after delivery
  APGAR scores in numerical values

CONTACTS AND LOCATIONS:
Overall Officials: Şerif Aksin, Assoc.Prof, Study Director — Siirt University Medical Faculty Obstetrics and Gynecology Departmant
Locations (1):
- Siirt Üniversity Medical Faculty, Siirt, Turkey (Türkiye)

REFERENCES:
- [Background] Vachon-Marceau C, Demers S, Markey S, Okun N, Girard M, Kingdom J, Bujold E. First-trimester placental thickness and the risk of preeclampsia or SGA. Placenta. 2017 Sep;57:123-128. doi: 10.1016/j.placenta.2017.06.016. Epub 2017 Jun 17. PMID 28864000
- [Background] Effendi M, Demers S, Giguere Y, Forest JC, Brassard N, Girard M, Gouin K, Bujold E. Association between first-trimester placental volume and birth weight. Placenta. 2014 Feb;35(2):99-102. doi: 10.1016/j.placenta.2013.11.015. Epub 2013 Dec 3. PMID 24345759
- [Background] Farina A. Systematic review on first trimester three-dimensional placental volumetry predicting small for gestational age infants. Prenat Diagn. 2016 Feb;36(2):135-41. doi: 10.1002/pd.4754. Epub 2016 Jan 19. PMID 26618611